CLINICAL TRIAL: NCT00310427
Title: NK1 Receptor Antagonism for Treatment of Anxiety and Craving in Anxious Alcohol Dependent Subjects During Early Abstinence
Brief Title: Effect of LY686017 on Alcohol Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Markus A. Heilig, M.D./National Institute on Alcohol Abuse and Alcoholism, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060129; 06-AA-0129; NCT00401037 (obsolete NCT alias)
Record Dates: First submitted 2006-04-01; First posted 2006-04-03 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Alcohol Dependence; Alcoholism
Keywords: Anxiety; Alcohol Dependence; Alcoholism
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — LY686017

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY686017 (Experimental): Subjects received 50 mg of the NK1 antagonist LY686017 orally on a daily basis.
  Interventions: Drug: LY686017
- Placebo (Placebo Comparator): Subjects received placebo orally on a daily basis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY686017 — 50 mg administered orally on a daily basis
  Arms: LY686017
Drug: Placebo — Administered on a daily basis
  Arms: Placebo

SUMMARY:
This study will determine whether the experimental drug LY686017 can reduce a person's desire for alcohol. A brain chemical called Substance P acts at places in the brain called NK1 receptors. Substance P is released in response to stress and gives rise to behaviors that are thought to represent anxiety. LY686017 blocks Substance P from acting at the NK1 receptors.

People between 21 and 65 years of age who have been drinking on a regular basis for at least one month before entering the study, who meet the criteria for alcohol dependence and who have an elevated score on a general test of anxiety may be eligible for this study.

Participants are admitted to the NIH Clinical Center for 35 days. They participate in an alcohol treatment program in addition to the research study. After having been withdrawn from alcohol for at least 2 days, participants receive either 50 mg of LY686017 or placebo (an inactive substance that looks like the study drug) every morning for 28 days. In addition to drug treatment, they undergo the following procedures:

* Functional magnetic resonance imaging (fMRI): In the last week of the study, subjects undergo MRI to study the amount of blood going to brain structures thought to be involved in anxiety and craving. During the procedure, they look at pictures of faces exhibiting various emotions and pictures related to alcohol.
* Cue reactivity: At the beginning and towards the end of the study, subjects are asked to rate their alcohol craving and their anxiety level while they sniff and handle their favorite alcoholic beverage or water.
* Metyrapone test: During weeks 1 and 4 of the study, subjects are given metyrapone - a drug that interferes with the body's ability to make the stress hormone cortisol - to determine how LY686017 affects the body's hormonal response. The drop in cortisol from metyrapone administration causes the brain to release ACTH, a hormone that causes the adrenal gland to make cortisol.
* Trier test: In the last week of the study, subjects give a 5-minute speech to three people and are then asked to subtract numbers in their head. Then they are asked to rate their feelings and desire for alcohol on two rating scales. Blood is drawn from a saline lock at the beginning and end of the test to measure hormone levels.
* Rating scales: Subjects complete an Obsessive Drinking Scale weekly and an Alcohol Urge Questionnaire and Comprehensive Psychiatric Rating Scale twice a week.
* Blood tests: Blood samples are collected periodically to check blood chemistries, clotting time, and the amount of LY686017 in the blood.

DETAILED DESCRIPTION:
Background:

Alcoholism is a chronic relapsing disorder characterized by cycles of intoxication interspersed with phases of withdrawal and abstinence. Co-morbidity with depression and anxiety disorders is high. Even in absence of independent psychiatric co-morbidity, anxiety symptoms are almost invariably present during early as well as protracted abstinence, sensitized over repeated cycles of intoxication and withdrawal, and are correlated with craving for alcohol upon exposure to alcohol associated cues. This psychopathology is likely to maintain the dependent state since it has been shown that stress and negative affective states are major relapse triggering factors. Substance P, released in the amygdala in response to stress, acts at NK1 receptors as an important mediator of behavioral stress effects in experimental animals. Blockade of this receptor subtype represents a novel principle for anxiolytic like actions, which is well documented in animal models and has some supportive data in humans. Furthermore, decreased opiate reward following NK1 receptor inaction is indicated by the reports that deletion of the NK1 receptor decreases both conditioned place preference and self-administration of opiates, while a similar reduction of alcohol reward is suggested by preliminary data showing decreased voluntary intake of alcohol in NK1 null-mutants.

Aims:

The present study is aimed at providing an initial, exploratory evaluation of whether the NK1 receptor is a candidate target for treatment of alcohol dependence that would merit further clinical development in conventional, full-scale clinical trial designs. To evaluate this, the aim of the present study is to determine whether NK1 antagonism can beneficially affect, in anxious alcohol dependent subjects during early abstinence, surrogate variables correlated with clinical outcomes, i.e.

* reduce craving for alcohol, measured as baseline self-reported urges, or in response to presentation of alcohol associated cues
* reduce negative affect
* influence corresponding objective measures (brain fMRI responses to alcohol-associated cues and to fear stimuli, respectively; and endocrine stress responses).

This study will address this aim using a novel, orally bioavailable and brain penetrant NK1 antagonist. Positive data in this exploratory study would be the first of their kind, and provide a rationale for evaluating the NK1 antagonist for anti-craving / anti-dipsotropic and anti-anxiety actions in alcohol dependent subjects in a longer term, suggesting that it might aid relapse prevention.

Methods:

The study will be carried out in 50 subjects aged 21-65 years, with alcohol dependence as their primary complaint, and without other serious medical or psychiatric conditions. An additional inclusion criterion will be the presence or history of significant anxiety symptoms on self report. Subjects will be admitted to the NIAAA research inpatient unit at the NIH Clinical Center through a platform training and natural history protocol which provides basic assessments and standard withdrawal treatment if needed. Patients will enter into the present protocol once such treatment, if needed, is completed. The present protocol will be started with a 1 week single blind placebo lead-in. During this phase, a baseline alcohol cue-reactivity session will be carried out according to established procedures, and urges to drink will be assessed. Cue-responsive subjects only, appr. 70% of alcohol dependent inpatients, will be randomized to active treatment or placebo, and enter the active treatment phase. The active treatment arm will receive 50 mg once daily of LY686017by oral intake, while the placebo group will continue to receive placebo in a double-blind fashion. The duration of active treatment will be 3 weeks.

Patients will remain hospitalized throughout this protocol. During this period, no psychotropic medication will be allowed, and abstinence from alcohol and other drugs will be monitored. Measures of craving will be obtained using: 1) ratings completed twice a week on the established Alcohol Urge Questionnaire (AUQ); 2) assessments of urge to drink (at baseline and under medication) during an established cue reactivity paradigm during which each patient undergoes an invivo exposure to his or her preferred alcoholic beverage. The medicated cue reactivity session will follow immediately after the Trier Test, a social stress task that independently induces urges for alcohol (stress induced craving); and augments subsequent cue-induced urges (stress-potentiated cue induced craving); 3) weekly assessment of alcohol related cognitions using the Obsessive Drinking Scale (ODS), a pharmacologically validated subscale of the established Obsessive Compulsive Drinking Scale (OCDS). In addition, measures of anxiety and depression symptoms will be obtained twice-weekly using the Comprehensive Psychiatric Rating Scale (CPRS). During the last treatment week, subjects will undergo an fMRI scan using established paradigms to evoke emotional responses, and to evoke alcohol-cue associated responses, respectively. Psychophysiological measures will be obtained in conjunction with the scan. Blood draws will be carried out on the day of the scan to allow for analysis of plasma concentrations of the experimental drug. The neuroendocrine stress response will be probed, using the standard metyrapone challenge test, in unmedicated state following the baseline CR session, and then again under active treatment or placebo following the fMRI scan.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 21 - 65.
* DSM-IV diagnosis of alcohol dependence on SCID, alcohol problems as primary complaint among substance use disorder, and alcohol use within the last month.
* Spielberger trait anxiety score greater than 39.
* Females of childbearing potential must agree to use a reliable method of birth control during the study. Reliable methods of birth control include oral contraceptives or Norplant(Registered Trademark); barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices; a partner with a vasectomy; or abstinence from intercourse.

EXCLUSION CRITERIA:

Subjects will be excluded if they meet any of the criteria below. The criteria for enrollment will be followed explicitly. If a subject who does not meet enrollment criteria is inadvertently enrolled, that subject will be discontinued from the study and Eli Lilly will be contacted.

General exclusion criteria for the NIAAA intramural treatment program:

* People who present with complicated medical problems requiring intensive medical or diagnostic management, such as hypertensive emergency, serious GI bleeding, major organ or body system dysfunction such as decompensated liver disease, renal failure, myocardial ischemia, congestive heart failure or cerebrovascular disease, major endocrine problems such as uncontrolled diabetes, pancreatic or thyroid disease.
* People who are infected with the Human Immunodeficiency Virus (HIV).
* Serious neuro-psychiatric conditions which impair judgment or cognitive function to an extent that precludes them from providing informed consent or complying with treatment, such as psychotic illness or severe dementia (incompetent individuals).
* People who are unlikely or unable to complete the treatment program because they become or are likely to be incarcerated while on the protocol.
* People who are required to receive treatment by a court of law or who are involuntarily committed to treatment.
* People with uncontrolled hypertension

Study specific exclusion criteria:

* People who are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* People who are employees of Eli Lilly & Co.
* Treatment within the last 30 days with a drug [not including study drug] that has not received regulatory approval for any indication at the time of study entry.
* A history of seizures, other than documented febrile seizures
* Patients with clinically significant hepatobiliary disease (as evaluated by a trained hepatologist) will be excluded from the protocol
* Pregnancy or lactation (negative pregnancy test required)
* Regular use of psychotropic medication (antidepressant, lithium, antipsychotic, anxiolytic, antiepileptic) within last 4 weeks, with the exception of benzodiazepines administered within the NIAAA program as part of alcohol withdrawal treatment.
* Inability or unwillingness to participate in an fMRI scan, including presence of metallic objects in the body, or pronounced claustrophobia
* Hypopituitarism or reduced adrenal secretory activity because of the risk of precipitating acute adrenal failure with metyrapone.
* Porphyria because metyrapone may be porphyrinogenic based on data from in-vitro systems.
* Thyroid dysfunction, which may alter the response to metyrapone.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anton RF, Moak DH, Latham PK. The obsessive compulsive drinking scale: A new method of assessing outcome in alcoholism treatment studies. Arch Gen Psychiatry. 1996 Mar;53(3):225-31. doi: 10.1001/archpsyc.1996.01830030047008. PMID 8611059
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780
- [Background] Brownell KD, Marlatt GA, Lichtenstein E, Wilson GT. Understanding and preventing relapse. Am Psychol. 1986 Jul;41(7):765-82. doi: 10.1037//0003-066x.41.7.765. No abstract available. PMID 3527003
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2006-AA-0129.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 subjects were initially screened for the study by undergoing a baseline alcohol cue reactivity test. Eight subjects were assessed as non-reactive and excluded from the study. In addition, 2 subjects refused to participate, and 3 subjects were excluded for other reasons. Thus, 53 subjects were randomized to the two treatment arms.
Period: Overall Study
Arm/Group | LY686017 | Placebo
Started | 27 | 26
Completed | 25 | 25
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY686017 | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 21 | 16 | 37
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Craving for Alcohol (Spontaneous)
Description: Alcohol craving was measured using the Alcohol Urges Questionnaire (AUQ). This is a self-report rating scale, with scores ranging from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | 19.7 (2.3) | 19.1 (2.4)

2. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 1, During the First of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 1/Rating 1 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -4.59 (1.70) | -1.52 (2.92)

3. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 1, During the Second of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 1 Rating 2 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -5.72 (2.13) | -4.14 (2.30)

4. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 2, During the First of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 2 Rating 1 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -6.40 (2.10) | -2.43 (2.69)

5. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 2, During the Second of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 2 Rating 2 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -6.88 (2.10) | -4.32 (2.52)

6. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 3, During the First of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 3 Rating 1 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -7.84 (1.88) | -3.33 (3.24)

7. Primary Outcome: Change From Baseline in Spontaneous Alcohol Craving at Week 3, During the Second of Two Weekly Ratings.
Description: as for outcome 1
Time Frame: Week 3 Rating 2 minus baseline
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | -9.24 (2.14) | -7.44 (2.58)

8. Primary Outcome: Craving for Alcohol Evoked by Alcohol-cue Challenge
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | LY686017 | Placebo
Number analyzed (Participants) | 25 | 25
Units on a scale | 19.2 (2.18) | 23.2 (2.62)

ADVERSE EVENTS:
Arm/Group | LY686017 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 14/25 | 18/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LY686017 (N=25) | Placebo (N=25)
Abdominal cramps (Gastrointestinal disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dizziness (General disorders) | 3 | 2
Fatigue (General disorders) | 11 | 5
Flatulence (Gastrointestinal disorders) | 1 | 2
Headache (General disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 3 | 2
Rash or pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Xerostomia (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes